CLINICAL TRIAL: NCT03772353
Title: Pyrotinib, Dalpiciclib(SHR6390) and Endocrine Therapy in Subjects With Dual-receptor Positive(ER+/HER2+) Advanced Breast Cancer: a Multi-center Phase Ib/II Study
Brief Title: Pyrotinib, Dalpiciclib(SHR6390) and Endocrine Therapy in Subjects With Dual-receptor Positive(ER+/HER2+) Advanced Breast Cancer
Acronym: PLEASURABLE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xichun Hu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLEASURABLE
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: hormone receptor; HER2; pyrotinib; CDK4/6 inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — dalpiciclib; pyrotinib; Letrozole; Fulvestrant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dalpiciclib combined with Pyrotinib and Endocrine therapy (Experimental): Data from phase Ib showed the triplet of pyrotinib, SHR6390, and letrozole had an acceptable safety profile and encouraging efficacy, potentially offering a chemotherapy-sparing treatment option for patients with HER2-positive/HR-positive MBC. Based on DLTs and clinical efficacy, pyrotinib 320mg/d, SHR6390 125mg/d, and letrozole 2.5mg/d was declared as RP2D. The pharmacokinetic analysis had not yielded conclusive results and would involve more samples in phase II trial.
  Dalpiciclib combined with Pyrotinib and Endocrine therapy (treatment of physician's choice: letrozole or fulvestrant) ER+/HER2+ metastatic breast cancer patients eligible for first- or second-line treatment were enrolled to receive dalpiciclib combined with pyrotinib and endocrine therapy (treatment of physician's choice: letrozole or fulvestrant)
  Interventions: Drug: Dalpiciclib; Drug: Pyrotinib; Drug: Letrozole; Drug: Fulvestrant

INTERVENTIONS:
Drug: Dalpiciclib — Dalpiciclib (SHR6390) is a novel small molecule inhibitor specifically targeting the CDK4/6 pathway.
  Other Names: SHR6390
Drug: Pyrotinib — Pyrotinib, an irreversible pan-ErbB receptor tyrosine kinase inhibitor, showed promising anti-tumour activity and acceptable tolerability in patients with HER2+ metastatic breast cancer (MBC)
Drug: Letrozole — Letrozole, a third-generation aromatase inhibitor, is the principal drug used in the treatment of postmenopausal patients with both early- and advanced-stage endocrine-responsive breast cancer (BC).
Drug: Fulvestrant — Fulvestrant is a selective oestrogen receptor (ER) degrader used in postmenopausal women with hormone receptor-positive advanced breast cancer

SUMMARY:
This is a single-center Ib / II study of triple targeted drug combination (endocrine therapy，novel HER2-targeted small molecule inhibitor pyrotinib and CDK4/6 inhibitor dalpiciclib(SHR6390) ) as a first or second line of therapy in patients with relapsed/metastatic hormone receptor positive and HER2-positive breast cancer.

DETAILED DESCRIPTION:
This is a single-center, single arm, open-label, run-in phase Ib / roll-over phase II study of endocrine therapy in combination with novel human epidermal growth factor receptor-2(HER2)-targeted tyrosine kinase Inhibitor pyrotinib and cyclin-dependent kinase 4/6(CDK4/6) Inhibitor dalpiciclib(SHR6390) in subjects with hormone receptor(HR)+/HER2+ relapsed or metastatic breast cancer. The study will enroll natural postmenopausal women, or women who have undergone bilateral oophorectomy.The phase Ib part of the study will determine safety and tolerability of the combination of endocrine therapy, pyrotinib and dalpiciclib to define that appropriate dose of dalpiciclib for phase II.Data from phase Ib showed the triplet of pyrotinib, dalpiciclib, andendocrine therapy had an acceptable safety profile and encouraging efficacy, potentially offering a chemotherapy-sparing treatment option for patients with HER2-positive/HR-positive MBC.Once the recommended regimen has been identified, subjects with the selected tumor type will be enrolled into expansion cohorts for the purpose of assessing efficacy and safety of the combination treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily joined the study, signed informed consent, and had good compliance.
2. Postmenopausal or premenopausal perimenopausal female patients aged ≥ 18 years and ≤ 75 years old,Meet one of the following:

   * Previous bilateral oophorectomy, or age ≥ 60 years; or Age <60, natural postmenopausal state (defined as regular months for at least 12 consecutive months After spontaneous cessation and no other pathological or physiological reasons),E2 and FSH in menopause Post-level; or
   * Pre-menopausal or perimenopausal female patients can also be included, but must be willing to receive treatment with LHRH agonists;
3. Patients with HR+/HER2+ recurrent or metastatic breast cancer confirmed by histopathology

   * HER2 positivity is defined by standard of 3+ staining by immunohistochemical staining (IHC) or positive for in situ hybridization (ISH)
   * Estrogen receptor(ER) or Progesterone receptor(PR) positive is defined as the percentage of cells positive for ER or PR expression ≥ 1%
   * Local recurrence needs to be confirmed by the physician that is unresectable
4. At least one extracranial measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.
5. Prior treatment:

   * Previously received no more than 1 prior lines of systemic treatment with trastuzumab regimen for repetitive metastatic diabetes [including anti-HER2 ADC, subsequent meaning is the same]

     1. The early stage includes trastuzumab-containing regimen treatment， or trastuzumab-containing regimen that relapses more than 1 year after the end of adjuvant treatment, and subsequent treatment is included as the first-line anti-HER2 treatment;
     2. The first-line treatment fails with the trastuzumab-containing regimen, or the trastuzumab-containing regimen recurs during the adjuvant treatment or relapses within 1 year after the adjuvant treatment ends, the follow-up treatment will be included as the second-line anti-HER2 treatment;
   * Have not received anti-HER2 TKI treatment before or received but did not prove that the treatment failed;
   * Past endocrine therapy has not proven resistance to aromatase inhibitors (definition of resistance: recurrence during or within 1 year after treatment with adjuvant aromatase inhibitors, received aromatase inhibitors in the recurrence and metastasis stage and disease progression), follow-up Letrozole is selected for endocrine therapy. Past endocrine therapy has aromatase inhibitor resistance, and follow-up endocrine therapy is fulvestrant.
6. Eastern Cooperative Oncology Group Performance Status of 0-1.
7. Life expectancy ≥ 12 weeks.
8. Adequate function of major organs meets the following requirements (no blood components and cell growth factors have been used within 14 days before randomization):

   * Neutrophils ≥ 1.5×10^9/L
   * Platelets ≥ 90×10^9/L
   * Hemoglobin ≥ 90g/L
   * Total bilirubin≤ 1.5 × the upper limit of normal (ULN)
   * ALT and AST ≤ 2.5 × ULN
   * BUN and Cr ≤ 1.5 × ULN
   * Left ventricular ejection fraction (LVEF) ≥ 50%
   * QTcF(Fridericia correction) ≤ 470 ms
   * International normalized ratio(INR)≤1.5 × ULN，activated partial thromboplastin time(APTT) ≤ 1.5 × ULN

Exclusion Criteria:

1. Meningeal metastasis or active brain parenchymal metastasis. Patients with clinically stable brain parenchymal metastases can be included, including asymptomatic brain metastases that have not received local treatment; or patients who have previously received central nervous system metastasis therapy (radiotherapy or surgery), if imaging confirms that stability has been maintained for at least 4 weeks , and have stopped symptomatic treatment (including hormones and mannitol, etc.) for more than 2 weeks
2. Previously received any CDK4/6 inhibitor treatment.
3. There are ascites, pleural effusion, pericardial effusion with clinical symptoms at baseline, those who need drainage, or those who have undergone drainage of serous effusion within 4 weeks before the first dose.
4. Inability to swallow, intestinal obstruction or other factors affecting the administration and absorption of the drug.
5. Received systemic therapy such as chemotherapy, molecular targeted therapy or other clinical trial drugs within 4 weeks before enrollment; received endocrine therapy within 2 weeks before enrollment.
6. Patients with other malignant tumors within 5 years or at the same time( except for cured skin basal cell carcinoma and cervical carcinoma in situ).
7. Have undergone major surgical procedures or significant trauma within 4 weeks prior to randomization, or are expected to undergo major surgery.
8. Pregnant women, lactating female, or women of childbearing age who are unwilling to take effective contraceptive measures.
9. Have a history of allergies to the drug components of this regimen.
10. Patients with active HBV and HCV infection; stable hepatitis B after drug treatment (HBV virus copy number is higher than the upper limit of reference value) and cured hepatitis C patients (HCV virus copy number exceeds the lower limit of detection method).
11. History of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency disease, history of organ transplantation.
12. History of cardiac dysfunction, include(1)angina (2)clinical significant arrythmia or require drug intervention (3)myocardial infarction (4)heart failure (5) other cardiac dysfunction (judged by the physician); any cardiac or nephric abnormal ≥ grade 2 found in screening.
13. Female patients who are pregnancy, lactation or women who are of childbearing potential tested positive in baseline pregnancy test.
14. Childbearing female who refuse to accept any contraception practice.
15. Determined by the physician, any serious coexisting disease might be harmful to the patient's safety or avoid the patients from accomplishing the treatment(e.g serious hypertension, diabetes, thyroid dysfunction,active infection etc.).
16. History of neurological or psychiatric disorders, including epilepsy or dementia.
17. Severe infections within 4 weeks prior to first dose (eg, intravenous infusion of antibiotics, antifungal or antiviral drugs according to clinical protocols), or unexplained fever (T > 38.3 °C ) during screening or prior to first administration.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-05-12 (Actual); Primary Completion 2023-06-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
The number of patients in the Phase 1b part of the study with any adverse events (AE). | 2 years
  To measure safety and tolerability of SHR6390 used in combination with and letrozole and pyrotinib (phase Ib part) we will assess the incidence, nature and severity of all adverse events (AE) that occur on or after C1D1 of therapy, AE severities will be classified using the CTCAE criteria.
Objective response rate (ORR) | 12 months
  According to recist1.1 standard, the proportion of patients whose best remission was CR or PR accounted for the total number of evaluable patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

REFERENCES:
- [Derived] Zhang J, Meng Y, Wang B, Wu X, Zheng H, Hu J, Liu W, Chen W, Wang L, Cao J, Tao Z, Li T, Ni S, Yu Z, Sun L, Wang Y, Peng Q, Wang S, Hu X, Wang J, Wu Y, Hu X. Dalpiciclib combined with pyrotinib and endocrine therapy in women with ER-positive, HER2-positive advanced breast cancer: A prospective, multicenter, single-arm, phase 2 trial. PLoS Med. 2025 Jul 31;22(7):e1004669. doi: 10.1371/journal.pmed.1004669. eCollection 2025 Jul. PMID 40743286
- [Derived] Zhang J, Meng Y, Wang B, Wang L, Cao J, Tao Z, Li T, Yao W, Hu X. Dalpiciclib Combined With Pyrotinib and Letrozole in Women With HER2-Positive, Hormone Receptor-Positive Metastatic Breast Cancer (LORDSHIPS): A Phase Ib Study. Front Oncol. 2022 Mar 7;12:775081. doi: 10.3389/fonc.2022.775081. eCollection 2022. PMID 35321427